CLINICAL TRIAL: NCT02347722
Title: Evaluation of Existing Biomarker Candidates to Accurately Classify the Etiology of Heart Failure
Brief Title: Biomarkers to Classify Heart Failure
Status: Active, not recruiting | Type: Observational
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Genome Canada (Other); Roche Diagnostics GmbH (Industry)
Responsible Party: Principal Investigator, Peter Liu, Chief Scientific Officer and VP of Research, Ottawa Heart Institute Research Corporation
Other Study IDs: 2014869-01H
Record Dates: First submitted 2015-01-21; First posted 2015-01-27 (Estimated); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure
Keywords: biomarkers; diagnosis; etiology of heart failure
MeSH Terms: conditions — Heart Failure; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Serum and plasma for biomarkers
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Retrospective: Heart failure patients where the etiology of their heart failure has been diagnosed. This cohort will consist of 3 groups: 1) Ischemic cardiomyopathy, 2) dilated cardiomyopathy and 3) diastolic heart failure
- Prospective: This cohort will consist of symptomatic heart failure patients diagnosed within 2 years.
- Healthy volunteers: Age matched healthy volunteers for comparison with heart failure patients

SUMMARY:
The purpose of this study is to evaluate existing biomarkers and see if they can be used to accurately diagnose the etiology of heart failure.

DETAILED DESCRIPTION:
This is a cohort study consisting of 2 patient cohorts. The first cohort will be studied retrospectively, using existing blood samples from different biobanks. Biomarkers will be measured and matched with the etiology of previously diagnosed heart failure by a biomarker panel of heart failure experts. This cohort consists of 100 patients each with (1) ischemic cardiomyopathy, (2) dilated cardiomyopathy and (3) diastolic heart failure. Blood samples will be analyzed for novel biomarkers. Investigators will be seeking biomarker candidate(s) alone or in combination which can predict each category of heart failure etiology with over 85% accuracy and the lowest levels of reclassification. A panel of heart failure experts will be assembled, and the appropriate cut-off values determined. Once this goal has been achieved, the prospective study will go ahead.

In the second cohort, biomarkers will be measured and used to diagnose the etiology of heart failure for each subject. This diagnosis will then be compared to the diagnosis from results of the usual diagnostic tests. Investigators will recruit 450 patients admitted to hospital or outpatient clinics with recently diagnosed heart failure (<2 years) and test for different biomarkers. Using the biomarker values, investigators will predict their heart failure etiology in an objective manner. The patients will then undergo definitive etiological workup as usual to establish the actual etiology of the heart failure. The duration of a typical etiological workup is about 3 days for hospitalized patients and up to 8 weeks for patients admitted to outpatient clinics. The predictive accuracy of the new heart failure panel will be compared to clinical assessment.

Investigators will perform cost-modeling in terms of the potential savings in avoiding unnecessary coronary angiographies or perfusion scans in a typical mixed cohort of heart failure patients based on the marker determined etiology.

A group of healthy volunteers will be added. This group will serve as age matched controls to the prospective cohort of heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted with symptomatic heart failure, diagnosed within 2 years.
* Diagnosis of congestive heart failure using the modified Framingham criteria:

Simultaneous presence of at least 2 major criteria or 1 major criterion in conjunction with 2 minor criteria or a previous clear diagnosis of heart failure.

Major criteria:

* Paroxysmal nocturnal dyspnea or orthopnea
* Neck vein distention
* Rales/Crackles (>10 cm from base of lungs)
* Acute pulmonary edema
* S3 gallop
* Increased central venous pressure (>16 cm H2O at right atrium)
* Hepatojugular reflux
* Weight loss >4.5 kg in 5 days in response to treatment Echocardiographic left ventricular dysfunction

Minor criteria:

* Bilateral ankle edema
* Nocturnal cough
* Dyspnea on exertion
* Hepatomegaly
* Pleural effusion
* Weight loss >4.5 kg caused by heart failure where factors other than treatment of CHF could have contributed to the weight loss
* Tachycardia (heart rate >120 beats/min) Minor criteria are acceptable only if they cannot be attributed to another medical condition (such as pulmonary hypertension, chronic lung disease, cirrhosis, ascites, or the nephrotic syndrome).

Exclusion Criteria:

* Patients unable to provide blood sample
* Patients unable to provide consent
* Patient with life expectancy of less than 6 months, or has major co-morbidities.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Participants who have participated in another research trial involving an investigational product in the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The retrospective cohort consists of stored blood samples from various biobanks.
  The prospective cohort consists of patients admitted to academic hospitals or outpatient clinics with symptomatic heart failure diagnosed within 2 years.
  The volunteer cohort consists of age matched healthy volunteers
Sampling Method: Probability Sample
Enrollment: 511 (Actual)
Dates: Start 2015-05; Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of heart failure panel to predict etiology of heart failure using biomarkers. | at end of study

SECONDARY OUTCOMES:
cost savings | At end of study

CONTACTS AND LOCATIONS:
Overall Officials: Peter Liu, MSc, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Data will be presented as the mean and standard deviation for the main cohort and sub-groups.